CLINICAL TRIAL: NCT00054665
Title: PS-341 and PS-341 + Epoch Chemotherapy and Molecular Profiling in Relapsed or Refractory Diffuse Large B-Cell Lymphomas
Brief Title: PS-341 Alone and PS-341 Plus EPOCH Chemotherapy to Treat Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Wyndham Wilson, Dr. Wyndham Wilson, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030096; 03-C-0096; NCT00057902 (obsolete NCT alias)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Results first posted 2012-09-11 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-08

CONDITIONS: B-Cell Lymphoma
Keywords: BCL-2; NFK-B; Drug Resistance; Translational; Lymphoma; Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma | interventions — Bortezomib; Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Prednisone; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: PS-341 Alone (Experimental): 1.3 mg/m^2 intravenous injection days 1, 4, 8, 11 every 3 weeks
  Interventions: Drug: PS-341
- Part B: PS-341 & EPOCH (Experimental): PS-341: level 1: 0.5 mg/m^2 intravenous (IV) days 1, 4; level 2: 1.0 mg/m^2 IV days 1, 4; level 3: 1.5 mg/m^2 IV days 1, 4; level 4: 1.7 mg/m^2 IV days 1, 4.
  EPOCH: Etoposide: 50 mg/m^2 day continuous intravenous infusion (CIV) days 1-4, 96 hour infusion; Doxorubicin: 10 mg/m^2 day CIV days 1-4, 96 hour infusion; Vincristine: 0.4 mg/m^2 day CIV days 1-4, 96 hour infusion; Cyclophosphamide: 750 mg/m^2 day IV day 5 bolus; Prednisone: 60 mg/m^2 by mouth twice a day days 1-5; Filgrastim: 300 micrograms subcutaneously days 6 to absolute neutrophil count recovery greater than or equal to 5000/mm^3. Repeat cycles every 21 days.
  Interventions: Drug: PS-341; Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Prednisone; Drug: Filgrastim

INTERVENTIONS:
Drug: PS-341 — 1.3 mg/m^2 intravenous injection days 1, 4, 8, 11 every 3 weeks
  Other Names: Velcade; Bortezomib; LDB-341; MLN-341
Drug: Etoposide — 50 mg/m^2 day continuous intravenous infusion (CIV) days 1-4, 96 hour infusion. Repeat cycle every 21 days.
  Other Names: Vepesid; VP-16
  Arms: Part B: PS-341 & EPOCH
Drug: Doxorubicin — 10 mg/m^2 day CIV days 1-4, 96 hour infusion. Repeat cycle every 21 days.
  Other Names: Adriamycin
  Arms: Part B: PS-341 & EPOCH
Drug: Vincristine — 0.4 mg/m^2 day CIV days 1-4, 96 hour infusion. Repeat cycle every 21 days.
  Other Names: Oncovin
  Arms: Part B: PS-341 & EPOCH
Drug: Cyclophosphamide — 750 mg/m^2 day IV day 5 bolus. Repeat cycle every 21 days.
  Other Names: Cytoxan
  Arms: Part B: PS-341 & EPOCH
Drug: Prednisone — 60 mg/m^2 by mouth twice a day days 1-5. Repeat cycle every 21 days.
  Other Names: Deltasone
  Arms: Part B: PS-341 & EPOCH
Drug: Filgrastim — 300 micrograms subcutaneously days 6 to absolute neutrophil count recovery greater than or equal to 5000/mm^3. Repeat cycle every 21 days.
  Other Names: Neupogen
  Arms: Part B: PS-341 & EPOCH

SUMMARY:
This study will examine the safety and effectiveness of an experimental drug called Bortezomib (PS-341), given alone and in combination with a chemotherapy regimen called Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin and Filgrastim (EPOCH), in treating non-Hodgkin's B-cell lymphoma. In the laboratory, PS-341 kills lymphoma cells and makes them more sensitive to chemotherapy. The EPOCH treatment regimen includes the drugs doxorubicin, etoposide, vincristine, cyclophosphamide, prednisone, and filgrastim.

Patients 18 years of age and older with an aggressive non-Hodgkin's lymphoma that has relapsed after treatment or is not responding to chemotherapy may be eligible for this study. Candidates will be screened with a medical history and physical examination. Other tests that may be required include blood and urine tests; lung function studies; imaging tests such as magnetic resonance imaging, computed tomography and x-rays; and biopsy (surgical removal of a small tissue sample) of tumor, bone marrow, or other tissue.

Upon entering the study, all participants will receive PS-341. The drug is given as a 3- to 5-second intravenous (through a vein) injection twice a week for 2 weeks. This is followed by a 1-week rest. Each 3-week period comprises one treatment cycle. The number of cycles a patient receives depends on how well he or she responds to the drug. Patients who do not have a complete remission or whose tumor grows on this therapy will be offered PS-341 in combination with up to six cycles of EPOCH chemotherapy. The treatment for patients taking PS-341 plus EPOCH is as follows:

* PS-341, given by 3- to 5-second intravenous (IV) injection on days 1 and 4 of each cycle.
* Doxorubicin, etoposide, and vincristine, given by continuous IV infusion over 4 days, beginning on day 1 and ending on day 5 of each cycle. The drugs are delivered through a lightweight portable infusion pump to an indwelling IV catheter (plastic tube) in a vein.
* Cyclophosphamide, given by IV infusion over 15 minutes on day 5 of each cycle.
* Prednisone, given by mouth (pills) twice a day on days 1 through 5 of each cycle.
* Filgrastim, given by injection under the skin starting on day 6 of each cycle and continuing until the white blood cell count increases or until day 19 of the cycle.

Patients also take a combination of antibiotics 3 days a week during EPOCH to prevent infection while resistance is lowered because of the chemotherapy. Etoposide, doxorubicin, and cyclophosphamide doses are adjusted as needed, based on white blood cell counts of the previous cycle. The first patients in the study will receive a low dose of PS-341. The dose will be increased in subsequent small groups of patients as long as the preceding dose is well tolerated.

Drug therapy for patients who are candidates for bone marrow transplant will be tailored to permit transplantation. Patients who are not eligible for or who choose not to have a bone marrow transplant will be followed at the National Institutes of Health (NIH) every 3 months the first year, every 4 months the second year, every 6 months the third year, and then once a year until their disease progresses or the study ends. Patients may have tumor and bone marrow biopsies, blood draws, and computed tomography (CT) scans periodically to evaluate disease status and drug side effects.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphomas (DLBCL) have been molecularly sub-classified into germinal center like B-cell (GCB) and activated B-cell like (ABC) DLBCL. Clinically, the ABC subtype has a significantly higher rate of drug resistance and lower survival. The ABC subtype has overexpression of nuclear factor-kappa B (NF-kB) with transcriptional activation of B cell lymphoma 2 (bcl-2), which may account for the drug resistance. The ability of NF-kB to inhibit responses to cancer therapeutic agents may also contribute to the refractory clinical behavior of ABC subtype, and inhibition of NF-kB can synergize with the chemotherapy to kill tumor cells. This protocol aims to study the affect of NF-kB inhibition, through proteasome inhibition by PS-341, on response to PS-341 and PS-341 with EPOCH chemotherapy in DLBCL. It will also assess the affect of PS-341 on NF-kB and BCL-2 tumor expression by microarray, and provide information on the specificity of PS-341.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Large B-cell lymphoma (subtypes: DLBCL (diffuse large B-cell lymphoma);

mediastinal (thymic) large B-cell lymphoma;

transformed large B-cell lymphoma;

follicular grade IIIB large B-cell lymphoma;

intravascular large B-cell lymphoma).

Confirmed pathological diagnosis at the treating institution.

Prior anthracycline-based treatment.

Age greater than or equal to 18 years.

Available tumor tissue for biopsy.

Eastern Cooperative Oncology Group (ECOG) performance 2 or better.

Major organ function: Absolute neutrophil count (ANC) greater than or equal to 1,000/microliters,

Platelet greater than or equal to 50,000/microliters,

creatinine less than or equal to 1.5 mg/dl or creatinine clearance greater than 60 cc/min;

serum glutamic pyruvic transaminase (SGPT) less than 5 x upper limit of normal;

bilirubin less than 2 mg/dl (total) except less than 5 mg/dl in patients with Gilbert's syndrome as defined by greater than 80 percent unconjugated; unless impairment due to organ involvement by lymphoma.

Informed consent and willingness to use contraception by both men and women.

Not pregnant or nursing because of an unknown potential for teratogenic or abortifacient effects.

Both male and female patients must be willing to use adequate contraception.

Human immunodeficiency virus (HIV) serology negative.

HIV positive patients receiving combination anti-retroviral therapy are excluded from the study because of positive pharmacokinetic interactions with PS-341 or the combination of PS-341 and EPOCH.

Additionally, the biology of HIV associated DLBCL's is often quite different from HIV negative disease due to involvement of Epstein Barr Virus (EBV).

Hepatitis B surface antigen negative.

No symptomatic cardiac disease or cardiac ejection fraction less than 40 percent (in patients receiving EPOCH).

No active central nervous system (CNS) lymphoma.

No systemic cytotoxic or experimental treatments within 4 weeks of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-02; Primary Completion 2008-09 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham Wilson, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (2):
- United States (2):
  - National Cancer Institute (NCI), Bethesda, Maryland
  - Roswell Parck Cancer Institute, Buffalo, New York

REFERENCES:
- [Background] Baldwin AS Jr. The NF-kappa B and I kappa B proteins: new discoveries and insights. Annu Rev Immunol. 1996;14:649-83. doi: 10.1146/annurev.immunol.14.1.649. PMID 8717528
- [Background] Dunleavy K, Pittaluga S, Czuczman MS, Dave SS, Wright G, Grant N, Shovlin M, Jaffe ES, Janik JE, Staudt LM, Wilson WH. Differential efficacy of bortezomib plus chemotherapy within molecular subtypes of diffuse large B-cell lymphoma. Blood. 2009 Jun 11;113(24):6069-76. doi: 10.1182/blood-2009-01-199679. Epub 2009 Apr 20. PMID 19380866
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2003-C-0096.html
- See also: CTCv2.0 — http://ctep.cancer.gov

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient was deemed ineligible and did not receive any treatment. In addition, per the protocol, patients who require an immediate treatment response for medical reasons will only receive part B of the protocol. This decision will be made by the principal investigator in consultation with the associate investigators (e.g. participants can skip A)
Groups:
- Part A: PS-341 Alone: 1.3 mg/m^2 intravenous bolus injection over 3-5 seconds every 3 weeks.Per the protocol, patients who require an immediate treatment response for medical reasons will only receive part B of the protocol. This decision will be made by the principal investigator in consultation with the associate investigators.
- Part B: PS-341 & EPOCH: PS-341 1.3 mg/m^2 intravenous bolus injection over 3-5 seconds every 3 weeks. EPOCH (etoposide 50 mg/m^2 day continuous intravenous infusion days 1-4, doxorubicin 10 mg/m^2 day continuous intravenous infusion days 1-4, vincristine 0.4 mg/m^2/day continuous intravenous infusion days 1-4, cyclophosphamide 750 mg/m^2 intravenous bolus day 5, prednisone 60 mg/m^2 by mouth days 1-5, and filgrastim 300 micrograms subcutaneously day 6 to absolute neutrophil count (ANC) recovery >/= 5000/mm^3.Per the protocol, patients who require an immediate treatment response for medical reasons will only receive part B of the protocol. This decision will be made by the principal investigator in consultation with the associate investigators.
Period: Part A
Arm/Group | Part A: PS-341 Alone | Part B: PS-341 & EPOCH
Started | 23 (5 participants only received Part A and 18 participants received Part B after Part A.) | 0
Completed | 23 | 0
Not Completed | 0 | 0
Period: Part B
Arm/Group | Part A: PS-341 Alone | Part B: PS-341 & EPOCH
Started | 0 | 44 (26 participants received only Part B)
Completed | 0 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A & B: PS-341 and PS-341 & EPOCH: Part A: PS-341 Alone
  1.3 mg/m^2 intravenous injection days 1, 4, 8, 11 every 3 weeks Part B: PS-341 & EPOCH
  PS-341: level 1: 0.5 mg/m^2 intravenous (IV) days 1, 4; level 2: 1.0 mg/m^2 IV days 1, 4; level 3: 1.5 mg/m^2 IV days 1, 4; level 4: 1.7 mg/m^2 IV days 1, 4.
  EPOCH: Etoposide: 50 mg/m^2 day continuous intravenous infusion (CIV) days 1-4, 96 hour infusion; Doxorubicin: 10 mg/m^2 day CIV days 1-4, 96 hour infusion; Vincristine: 0.4 mg/m^2 day CIV days 1-4, 96 hour infusion; Cyclophosphamide: 750 mg/m^2 day IV day 5 bolus; Prednisone: 60 mg/m^2 by mouth twice a day days 1-5; Filgrastim: 300 micrograms subcutaneously days 6 to absolute neutrophil count recovery greater than or equal to 5000/mm^3. Repeat cycles every 21 days
Arm/Group | Arm A & B: PS-341 and PS-341 & EPOCH
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 53.04 (16.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 45
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate
Description: Clinical Response Rate is the number of participants with a partial and complete response assessed by the criteria for lymphoma. A complete response is complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy and normalization of those biochemical abnormalities. Partial response is a greater than or equal to 50% decrease in the sum of the products of the greatest diameters of 6 largest dominant nodes or nodal masses. No increase in size of nodes, liver or spleen and no new sites of disease
Time Frame: 18 weeks
Measure: Number; unit: Participants
Groups:
- Part B: PS-341 & EPOCH: PS-341: level 1: 0.5 mg/m^2 intravenous (IV) days 1, 4; level 2: 1.0 mg/m^2 IV days 1, 4; level 3: 1.5 mg/m^2 IV days 1, 4; level 4: 1.7 mg/m^2 IV days 1, 4.
  EPOCH: Etoposide: 50 mg/m^2 day continuous intravenous infusion (CIV) days 1-4, 96 hour infusion; Doxorubicin: 10 mg/m^2 day CIV days 1-4, 96 hour infusion; Vincristine: 0.4 mg/m^2 day CIV days 1-4, 96 hour infusion; Cyclophosphamide: 750 mg/m^2 day IV day 5 bolus; Prednisone: 60 mg/m^2 by mouth twice a day days 1-5; Filgrastim: 300 micrograms subcutaneously days 6 to absolute neutrophil count recovery greater than or equal to 5000/mm^3. Repeat cycle every 21 days.
Arm/Group | Part A: PS-341 Alone | Part B: PS-341 & EPOCH
Number analyzed (Participants) | 23 | 44
Participants
  Partial response | 1 | 7
  Complete response | 0 | 8

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 43 months
Measure: Number; unit: Participants
Groups:
- Part A: PS-341 Alone: Part A: 1.3 mg/m^2 intravenous injection days 1, 4, 8, 11 every 3 weeks
- Part B: PS-341 & EPOCH: Part B:
  PS-341: level 1: 0.5 mg/m^2 intravenous (IV) days 1, 4; level 2: 1.0 mg/m^2 IV days 1, 4; level 3: 1.5 mg/m^2 IV days 1, 4; level 4: 1.7 mg/m^2 IV days 1, 4.
  EPOCH: Etoposide: 50 mg/m^2 day continuous intravenous infusion (CIV) days 1-4, 96 hour infusion; Doxorubicin: 10 mg/m^2 day CIV days 1-4, 96 hour infusion; Vincristine: 0.4 mg/m^2 day CIV days 1-4, 96 hour infusion; Cyclophosphamide: 750 mg/m^2 day IV day 5 bolus; Prednisone: 60 mg/m^2 by mouth twice a day days 1-5; Filgrastim: 300 micrograms subcutaneously days 6 to absolute neutrophil count recovery greater than or equal to 5000/mm^3. Repeat cycle every 21 days.
Arm/Group | Part A: PS-341 Alone | Part B: PS-341 & EPOCH
Number analyzed (Participants) | 23 | 44
Participants | 23 | 44

ADVERSE EVENTS:
Groups:
- Part A: PS-341 Alone: PS-341 1.3 mg/m^2 intravenous injection days 1, 4, 8, 11 every 3 weeks
Arm/Group | Part A: PS-341 Alone | Part B: PS-341 & EPOCH
Serious Adverse Events (participants affected / at risk) | 21/24 | 40/44
Other Adverse Events (participants affected / at risk) | 24/24 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: PS-341 Alone (N=24) | Part B: PS-341 & EPOCH (N=44)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 6 (18) | 17 (39)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 7 (8) | 17 (43)
Leukocytes (total WBC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 5 (8) | 13 (25)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5 (6) | 21 (41)
Platelets (Blood and lymphatic system disorders) | 12 (27) | 33 (80)
Transfusion: Platelets (Blood and lymphatic system disorders) | 1 (1) | 12 (22)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 1 (1) | 13 (19)
Vasovagal episode (Cardiac disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 1 (1) | 5 (6)
Hypotension (Cardiac disorders) | 4 (7) | 11 (13)
Partial thromboplastin time (PTT) (Investigations) | 3 (3) | 4 (5)
Prothrombin time (PT) (Investigations) | 1 (1) | 1 (1)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 8 (9) | 10 (14)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC< (General disorders) | 3 (3) | 3 (3)
Rigors, chills (General disorders) | 1 (1) | 0 (0)
Sweating (diaphoresis) (General disorders) | 1 (1) | 0 (0)
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Anorexia (Gastrointestinal disorders) | 4 (4) | 8 (8)
Constipation (Gastrointestinal disorders) | 1 (3) | 6 (6)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 7 (9) | 11 (16)
Nausea (Gastrointestinal disorders) | 7 (8) | 12 (17)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 2 (2) | 8 (14)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 3 (3) | 6 (6)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (7)
Alkaline phosphatase (Hepatobiliary disorders) | 1 (1) | 3 (5)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1) | 9 (11)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 2 (4) | 4 (5)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 3 (3) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 4 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 5 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 4 (6)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 4 (5)
Ataxia (incoordination) (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness/lightheadedness (Nervous system disorders) | 2 (3) | 4 (7)
Neuropathy - motor (Nervous system disorders) | 1 (1) | 2 (2)
Neuropathy-sensory (Nervous system disorders) | 5 (5) | 8 (10)
Syncope (fainting) (Nervous system disorders) | 1 (2) | 1 (1)
Ocular/Visual-Other (Specify, periorbital edema) (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain or cramping (Gastrointestinal disorders) | 3 (3) | 5 (6)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Neuropathic pain (Nervous system disorders) | 1 (4) | 1 (1) — (e.g., jaw pain, neurologic pain, phantom limb pain, post-infectious neuralgia, or painful neuropathies)
Inner ear/hearing (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Prolonged QTc interval (QTc > 0.48 seconds) (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (PVCs/bigeminy/trigeminy/ventricular tachycardia) (Cardiac disorders) | 0 (0) | 1 (1)
Weight loss (General disorders) | 0 (0) | 2 (2)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal-Other (Gastrointestinal disorders) | 0 (0) | 2 (2) — tongue swollen rectal incontinence
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Bilirubin (Hepatobiliary disorders) | 0 (0) | 3 (4)
Febrile neutropenia (Infections and infestations) | 0 (0) | 5 (6) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection (Infections and infestations) | 0 (0) | 9 (12) — (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e9/L)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 0 (0) | 7 (13)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Chest pain (non-cardiac and non-pleuritic) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain-Other (Specify, testicular) (General disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
Bicarbonate (Investigations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 10 (14)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Mood alteration-anxiety agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Neurology-Other (Specify) (Nervous system disorders) | 0 (0) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary-Other (Specify, wheezing) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Constitutional Symptoms-Other (Specify, generalized weakness) (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: PS-341 Alone (N=24) | Part B: PS-341 & EPOCH (N=44)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (1) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5) | 26 (40)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 5 (5) | 25 (48)
Lymphopenia (Blood and lymphatic system disorders) | 6 (8) | 14 (22)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (2) | 26 (46)
Platelets (Blood and lymphatic system disorders) | 4 (10) | 14 (26)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 1 (1) | 18 (21)
Edema (General disorders) | 6 (6) | 2 (3)
Phlebitis (superficial) (Cardiac disorders) | 1 (1) | 1 (1)
Prothrombin time (PT) (Investigations) | 1 (1) | 3 (5)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1) | 10 (12)
Fever (General disorders) | 3 (4) | 9 (11) — (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L)
Weight gain (General disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Anorexia (Gastrointestinal disorders) | 7 (7) | 7 (8)
Constipation (Gastrointestinal disorders) | 7 (7) | 9 (13)
Dehydration (Gastrointestinal disorders) | 1 (1) | 6 (7)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 3 (6) | 6 (6)
Dyspepsia/heartburn (Gastrointestinal disorders) | 2 (2) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 4 (4)
Mouth dryness (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4) | 13 (15)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 2 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (4) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hemorrhage-Other (Specify, L. eye) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Alkaline phosphatase (Hepatobiliary disorders) | 3 (3) | 4 (4)
Hypoalbuminemia (Hepatobiliary disorders) | 3 (4) | 21 (25)
Infection (documented clinically or microbiologically) with grade 3 or 4 (Infections and infestations) | 1 (1) | 7 (9)
Infection without neutropenia (Infections and infestations) | 5 (12) | 5 (6)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 0 (0)
Amylase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperglycemia (Hepatobiliary disorders) | 4 (6) | 15 (21)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 9 (13)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (5) | 16 (20)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 15 (24)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 14 (20)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 18 (24)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dizziness/lightheadedness (Nervous system disorders) | 1 (1) | 4 (4)
Insomnia (Nervous system disorders) | 2 (2) | 4 (4)
Neuropathy-sensory (Nervous system disorders) | 2 (2) | 12 (13)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal pain or cramping (Gastrointestinal disorders) | 6 (9) | 7 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 8 (8)
Chest pain (non-cardiac and non-pleuritic) (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 5 (6) | 12 (14)
Pain due to radiation (General disorders) | 1 (1) | 0 (0)
Pain-Other (Specify) (General disorders) | 1 (2) | 3 (3) — wisdom tooth testicular pain tooth pain low back
Pelvic pain (Reproductive system and breast disorders) | 2 (3) | 0 (0)
Tumor pain (onset or exacerbation of tumor pain due to treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dysuria (painful urination) (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Musculoskeletal-Other (Specify, degenerative changes-L. spine) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Transfusion: Platelets (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 4 (4)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 0 (0) | 2 (2)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 4 (5)
Pericardial effusion/pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Thrombosis/embolism (Cardiac disorders) | 0 (0) | 3 (3)
Partial thromboplastin time (PTT) (Investigations) | 0 (0) | 8 (8)
Constitutional Symptoms-Other (Specify, disease progression) (General disorders) | 0 (0) | 1 (1)
Rigors, chills (General disorders) | 0 (0) | 1 (1)
Sweating (diaphoresis) (General disorders) | 0 (0) | 2 (2)
Weight loss (General disorders) | 0 (0) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 0 (0) | 2 (2)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 0 (0) | 3 (5) — Abdominal bloating Abd. fullness Lost a filling on L. maxillary Tooth extraction
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 0 (0) | 19 (26)
Bilirubin (Hepatobiliary disorders) | 0 (0) | 7 (7)
SGOT (aspartate aminotransferase (AST)) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 0 (0) | 4 (4)
SGPT (alanine aminotransferase (ALT)) (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 9 (11)
Febrile neutropenia (Infections and infestations) | 0 (0) | 6 (7) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Bicarbonate (Investigations) | 0 (0) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 7 (8)
Lipase (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Mood alteration-depression (Psychiatric disorders) | 0 (0) | 1 (1)
Neurologic-Other (Specify) (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 2 (2)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (8)
Neuropathic pain (e.g. jaw pain, neurologic pain, phantom pain, limb pain, post-infectious neuralgi (Nervous system disorders) | 0 (0) | 2 (3)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 10 (11)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pulmonary-Other (Specify, wheezing) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Creatinine (Renal and urinary disorders) | 0 (0) | 6 (9)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No